CLINICAL TRIAL: NCT05349279
Title: Disease Registry for Pregnant Women With Suspected COVID-19 or Confirmed SARS-CoV-2 and Their Neonates.
Brief Title: Qatar PREgnancy Covid-19 OUtcome Study
Acronym: QPRECIOUS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hamad Medical Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: MRC-01-21-122
Record Dates: First submitted 2022-04-26; First posted 2022-04-27 (Actual); Last update posted 2022-05-20 (Actual); Status verified 2021-09

CONDITIONS: COVID-19; Pregnant Women
Keywords: Pregnant woman; COVID-19 infection; Postpartum women; Neonates
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The in-utero exposure of acute viral infection in some instances is proven to have short- and long-term neonatal effects during the postnatal and childhood period and the Zika virus, measles, mumps, and rubella are few examples. COVID-19 is caused by a novel coronavirus strain of unknown consequences. The main purpose of this registry is to collect baseline data and help to establish future studies and hypothesis generation.

In addition, we will be exploring the psychological impact of COVID-19 on women during the pregnancy and postnatal period. Stress and anxiety level are increased with potential adverse pregnancy and/or neonatal outcomes especially during an infectious disease outbreak. In fact, COVID-19 is associated with adverse maternal and neonatal outcomes resulting in increased levels of stress and anxiety. In addition, women during the pregnancy, peripartum, and postpartum period are at increased risk of depression. A risk that has been aggravated by social and physical isolation. Indeed, the social and physical isolation, a critically needed measure to stop the virus transmission, resulted in increased stress and depression levels and adversely affecting the mental and physical health of both the mother and the baby.

DETAILED DESCRIPTION:
The coronavirus disease 2019 or 'COVID-19' is a respiratory tract infection caused by the novel coronavirus strain initially (1). On 12th March 2020, the World Health Organization declared it as a 'pandemic' outbreak of utmost international concern. The majority of the published evidence has originated from China, where the first coronavirus patient was identified in Wuhan City in December 2019 (2,3). Previous emerging infections such as H1N1 influenza virus, Zika virus, severe acute respiratory syndrome coronavirus (SARS-CoV), and Middle East respiratory syndrome coronavirus (MERSCoV) have been shown to have a significant impact on maternal as well as perinatal outcomes (4,5).

The obstetrical population is considered vulnerable. Pregnancy involves multiple interactions with the health care system and eventually all are admitted to the hospital for delivery, therefore, managing the pregnant population presents a unique challenge during this pandemic. Additionally, the physiological changes and partial immune suppression during pregnancy make pregnant women and newborn babies susceptible to several infections. Post-partum hemorrhage, maternal sepsis, preeclampsia, premature rupture of the membrane are the most common adverse events reported to have been caused by this disease in pregnant women (11).

From the limited information gathered about the novel coronavirus, its impact on pregnancy and newborn, and the drastically increasing burden of the disease, it is vital that scientific information concerning the disease is collected and shared in a concise and practical manner. Hence, there is a need to collect case data rapidly, to pool global data on the natural history of women affected by suspected COVID-19 or confirmed SARS-CoV-2 in pregnancy to inform treatment and implement preventative strategies in this and future outbreaks. A center-based registry, gathering case data prospectively on the effect of SARS-CoV-2 infection from healthcare systems around the world offers a method to accrue clinical outcomes on key research questions from a variety of populations, and the Q- PRECIOS register will serve such purpose.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant woman with suspected or confirmed SARS-CoV-2 infection
* Postpartum women who delivered during the last six weeks and
* Neonate(s) of women included in the registry

Exclusion Criteria:

* Nonpregnant woman with suspected or confirmed SARS-CoV-2 infection
* Postpartum women who delivered after six weeks

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — The COVID-19 infection during pregnancy and postnatal period.
Study Population: We will include all pregnant patients with suspected or confirmed COVID-19 infection at all HMC facilities including WWRC, CH, AKH, AWH, and its associated quarantine sites and their offspring's
Sampling Method: Non-Probability Sample
Enrollment: 4000 (Estimated)
Dates: Start 2021-05-25 (Actual); Primary Completion 2023-04-15 (Estimated); Study Completion 2023-04-15 (Estimated)

PRIMARY OUTCOMES:
Retrospective Study | April 2021 - April 2023
  Prevalence of COVID-19 and its associated sign and symptoms in pregnancy in Qatar
Prospective Study | April 2021 - April 2023
  Maternal and neonatal demographic and outcomes pf pregnant women affect with COVID-19

CONTACTS AND LOCATIONS:
Overall Officials: Mahmoud Gasim Mohamed, M.SC, Study Director — Department of Pharmacy, Women's wellness and research center, Hamad Medical Corporatiom; Salwa Abo Yaqoub, MBBS, Principal Investigator — Hamad Medical Corporation
Locations (1):
- Women's Wellness and Research Center, Doha, Qatar

REFERENCES:
- [Result] (1) Sohrabi C, Alsafi Z, O'Neill N, Khan M, Kerwan A, Al-Jabir A, et al. World Health Organization declares global emergency: A review of the 2019 novel coronavirus (COVID-19). International Journal of Surgery. 2020 (2) World Health Organization. WHO Director-General's opening remarks at the media briefing on COVID-19-11 March 2020. Geneva, Switzerland. 2020;. (3) Guo Y, Cao Q, Hong Z, Tan Y, Chen S, Jin H, et al. The origin, transmission and clinical therapies on coronavirus disease 2019 (COVID-19) outbreak-an update on the status. Military Medical Research. 2020; 7(1):1-10. (4) Moore CA, Staples JE, Dobyns WB, Pessoa A, Ventura CV, Da Fonseca EB, et al. Characterizing the pattern of anomalies in congenital Zika syndrome for pediatric clinicians. JAMA pediatrics. 2017; 171(3):288-295. (5) Rasmussen SA, Jamieson DJ, Honein MA, Petersen LR. Zika virus and birth defects-reviewing the evidence for causality. New England Journal of Medicine. 2016; 374(20):1981-1987. (6) The World Health Organisation. Coronavirus disease (COVID-19) Pandemic. [homepage on the Internet]. World Health Organisation; 2020 [updated April/26; cited 2020 April/26]. Available from: https://www.who.int/emergencies/diseases/novel-coronavirus-2019. (7) Surveillances V. The epidemiological characteristics of an outbreak of 2019 novel coronavirus diseases (COVID-19)-China, 2020. China CDC Weekly. 2020; 2(8):113-122. (8) Adhikari SP, Meng S, Wu Y, Mao Y, Ye R, Wang Q, et al. Epidemiology, causes, clinical manifestation and diagnosis, prevention and control of coronavirus disease (COVID-19) during the early outbreak period: a scoping review. Infectious diseases of poverty. 2020; 9(1):1-12. (9) Lai C, Shih T, Ko W, Tang H, Hsueh P. Severe acute respiratory syndrome coronavirus 2 (SARS- CoV-2) and coronavirus disease-2019 (COVID-19): the epidemic and the challenges. International journal of antimicrobial agents. 2020; :105924. (10) Mullins E, Evans D, Viner R, O'Brien P, Morris E. Coronavirus in pregnancy and delivery: a rapid review. Ultrasound in Obstetrics & Gynecology. 2020;. (11) The Royal College of Obstetricians and Gynaecologists (RCOG). Coronavirus (COVID-19) Infection in Pregnancy. London, United Kingdom: Royal College of Obstetricians and Gynaecologists; 2020. (12) Alzamora MC, Paredes T, Caceres D, Webb CM, Valdez LM, La Rosa M. Severe COVID-19 during Pregnancy and Possible Vertical Transmission. American Journal of Perinatology. 2020;. (13) Karami P, Naghavi M, Feyzi A, Aghamohammadi M, Novin MS, Mobaien A, et al. Mortality of a pregnant patient diagnosed with COVID-19: A case report with clinical, radiological, and histopathological findings. Travel Medicine and Infectious Disease. 2020; :101665. (14) Liu Y, Chen H, Tang K, Guo Y. Clinical manifestations and outcome of SARS-CoV-2 infection during pregnancy. The Journal of infection. 2020;. (15) Chen H, Guo J, Wang C, Luo F, Yu X, Zhang W, et al. Clinical characteristics and intrauterine vertical transmission potential of COVID-19 infection in nine pregnant women: a retrospective review of medical records. The Lancet. 2020; 395(10226):809-815. (16) Wang1a X, Zhou2a Z, Zhang J, Zhu F, Tang Y, Shen X, et al. A case of 2019 Novel Coronavirus in a pregnant woman with preterm delivery. Clin Infect Dis. 2020; (17) Zhu H, Wang L, Fang C, Peng S, Zhang L, Chang G, et al. Clinical analysis of 10 neonates born to mothers with 2019-nCoV pneumonia. Translational pediatrics. 2020; 9(1):51.

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-11-04): https://cdn.clinicaltrials.gov/large-docs/79/NCT05349279/Prot_SAP_000.pdf
  • Informed Consent Form (2020-11-04): https://cdn.clinicaltrials.gov/large-docs/79/NCT05349279/ICF_001.pdf